CLINICAL TRIAL: NCT03635463
Title: Effect of Modified Twin Block in Skeletal Class II Growing Females With Mandibular Deficiency: A Randomized Controlled Trial
Brief Title: Effect of Modified Twin Block in Skeletal Class II Growing Females With Mandibular Deficiency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Heba Yehia, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-CU-2018-08-05
Record Dates: First submitted 2018-08-15; First posted 2018-08-17 (Actual); Last update posted 2018-12-03 (Actual); Status verified 2018-11

CONDITIONS: Class II Division 1 Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class II

STUDY DESIGN:
Who Masked: Participant
Masking Description: double blinded( participant and outcome assessor)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- twin block appliance (Experimental): this group will receive conventional twin block appliance and followed up every month for 9 months.
  Interventions: Device: twin block appliance
- modified twin block appliance group (Experimental): modified twin block appliance group , this group will receive the modified appliance and followed up every month for 9 months
  Interventions: Device: modified twin block appliance

INTERVENTIONS:
Device: twin block appliance — a functional appliance that enhances mandibular growth in growing patients made from vaccum sheets (esthetic)
  Other Names: mandibular functional appliance
  Arms: twin block appliance
Device: modified twin block appliance — a convetional twin block functional appliance that enhances mandibular growth in growing patients
  Arms: modified twin block appliance group

SUMMARY:
The aim of this study is to evaluate the treatment effects of conventional twin block appliance versus modified twin block appliance in the treatment of patients in growing stage having skeletal class II division 1 with mandibular deficiency.

DETAILED DESCRIPTION:
in this randomized controlled trail there are 2 groups , the first group will receive modified twin block appliance ,in the second group will receive conventional twin block appliance . the follow up period will be 9 months till mandibular growth occur . the assessment will be through a questionnaire on the number of hours the appliance is worn each day , and another questionnaire assessing the difficulty of speech and aesthetics . Also by, photographs, x-rays and study models preoperative and post operative.

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal Class II relationship (ANB > 4°).
2. Mandibular retrognathy (SNB < 78°).
3. Overjet ≥ 5 mm.
4. Minimal crowding in dental arches (≤4 mm).
5. Class II molar relation.
6. Growing female patients.
7. Patients with CMV3 maturation stage of the cervical verbrae.

Exclusion Criteria:

1. No history of orthodontic treatment either prior to or during functional Appliance therapy.
2. Posterior cross bites or severe maxillary transverse deficiency.
3. Severe facial asymmetry determined by clinical or radiographical examination.
4. Poor oral hygiene.
5. Systemic diseases that may affect the orthodontic treatment results.
6. Patients past their peak growth spurt.

Ages: 9 Years to 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
enhancing mandibular skeletal growth | 9 months
  it will be assessed by measuring the incremental growth by quick ceph (mm)

SECONDARY OUTCOMES:
dentoalveolar changes | 9 months
  quick ceph (mm)
Improvement of soft tissue profile | 9 months
  quick ceph (mm)
Patient's compliance | 9 months
  table chart (no of hours/day)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol